CLINICAL TRIAL: NCT01799148
Title: Impact of AIR Pollution on Inflammation, Oxidative Stress and 1-year Prognosis in Patients Hospitalized for Acute COronary Syndrome
Brief Title: Air Pollution, Inflammation and Acute Coronary Syndrome
Acronym: AIRACOS
Status: Completed | Type: Observational
Sponsor: Fundación Canaria Rafael Clavijo para la Investigación Biomédica (Other)
Responsible Party: Principal Investigator, Alberto Domínguez Rodríguez, Alberto Dominguez Rodriguez, Fundación Canaria Rafael Clavijo para la Investigación Biomédica
Other Study IDs: AIRACOS; AIRACOS-CANARY ISLANDS (Other: Hospital Universitario de Canarias)
Record Dates: First submitted 2013-02-23; First posted 2013-02-26 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Patients With Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Air pollution.; Inflammation.; Oxidative Stress.; Prognosis
MeSH Terms: conditions — Acute Coronary Syndrome; Inflammation | interventions — Particulate Matter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 360 Days

GROUPS / COHORTS (1):
- Particulate air pollutants: Cohort of consecutive patients admitted with diagnosis of acute coronary syndrome in the cardiology unit of a tertiary hospital, which will quantify the exposure of particulate air pollutants 24 hours a day 7 days earlier prior to admission.
  Interventions: Other: Particulate air pollutants

INTERVENTIONS:
Other: Particulate air pollutants — We will determined the average concentrations of different sizes of particulate matter from 1 day or up to 7 days prior to admission in patients with acute coronary syndrome.

SUMMARY:
The objectives of this study are: 1) To determine whether patients with acute coronary syndrome, the level of environmental exposure to particulate air pollutants in the week prior to admission, are related to concentrations of inflammatory molecules and oxidative stress. 2) To investigate whether the level of environmental exposure is an independent prognostic factor in terms of overall and cardiovascular mortality, myocardial infarction or unstable angina at 30 days, 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute coronary syndrome

Exclusion Criteria:

* Infectious process and / or local or systemic inflammation in the 15 days before admission.
* Thyrotoxicosis.
* Neoplasms - or any other disease that seriously compromise the prognosis of life and / or generate a systemic inflammatory response.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of consecutive patients admitted with diagnosis of aucte coronary, which will quantify the exposure of particulate air pollutants 24 hours a day 7 days earlier prior to admission. Also be determined inflammatory molecules and oxidative stress in admission. During the evolution of these patients, after 30 days, 6 and 12 months will recorded major adverse cardiovascular events. It also will quantify the exposure of air pollutant particles, in all patients included at 30 days, 6 and 12 months.
Sampling Method: Probability Sample
Enrollment: 307 (Actual)
Dates: Start 2011-11; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Impact of air pollution on inflammation, oxidative stress and 1-year prognosis in patients hospitalized for acute coronary syndrome. | 7 days
  A single center, cohort of consecutive patients admitted with diagnosis of acute coronary syndrome in the cardiology unit of a tertiary hospital, which will quantify the exposure of particulate air pollutants 24 hours a day 7 days earlier prior to admission. Also be determined inflammatory molecules and oxidative stress in admission.

SECONDARY OUTCOMES:
Impact of air pollution on inflammation, oxidative stress and 1-year prognosis in patients hospitalized for acute coronary syndrome. | 1 year
  During the evolution of these patients, after 30 days, 6 and 12 months will recorded major adverse cardiovascular events. It also will quantify the exposure of air pollutant particles in all patients included, at 30 days, 6 and 12 months.

OTHER OUTCOMES:
Impact of air pollution on inflammation, oxidative stress and 1-year prognosis in patients hospitalized for acute coronary syndrome: | 1 year
  During the evolution of these patients, after 30 days, 6 and 12 months will recorded major adverse cardiovascular events. It also will quantify the exposure of air pollutant particles in all patients included, at 30 days, 6 and 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain

REFERENCES:
- [Derived] Dominguez-Rodriguez A, Rodriguez S, Abreu-Gonzalez P, Avanzas P. [Impact of air pollution on inflammation, oxidative stress and 1-year prognosis in patients hospitalized for acute coronary syndrome: design of the AIRACOS study]. Med Clin (Barc). 2013 Dec 21;141(12):529-32. doi: 10.1016/j.medcli.2013.05.024. Epub 2013 Jul 25. No abstract available. Spanish. PMID 23891131